CLINICAL TRIAL: NCT01658059
Title: Reducing Children's Anxiety Using Homeopathic Remedy Before Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moti Moskovitz, clinical senior lecturer, department of pediatric dentistry, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: rcauhr-HMO-CTIL
Record Dates: First submitted 2012-07-21; First posted 2012-08-06 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Children's Dental Anxiety
MeSH Terms: interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Experimental): homeopathic remedy first , placebo second
  Interventions: Other: Homeopathic remedy; Other: Placebo
- group 2 (Experimental): placebo first, homeopathic remedy second
  Interventions: Other: Homeopathic remedy; Other: Placebo

INTERVENTIONS:
Other: Homeopathic remedy — drops of the homeopathic remedy will be taken twice a day before the treatment and once on the morning of the treatment day.
Other: Placebo — drops of the placebo will be taken twice a day before the treatment and once on the morning of the treatment day.

SUMMARY:
Pharmacological interventions to aid behavior management's techniques are commonly used in pediatric dentistry. The aim of the medicaments is to control behavior and allow safe completion of a dental procedure. Homeopathic remedy is safe and can be effective to control behavior and decrease anxiety in children during dental treatment.

Aim: 1. To explore the efficacy of homeopathic drugs in decreasing children's dental anxiety before dental treatment.

2. To assess the effectiveness of homeopathic remedy in facilitating dental treatment for anxious children.

Methods: prospective, double-blind study. Thirty healthy children (5-12 years-old) will receive homeopathic remedy\placebo before dental treatment. Anxiety reduction will be measured using: saliva cortisol levels, saliva α-amylase levels, facial image scale (FIS), and Houpt behavior scale.

Expected results: the homeopathic remedy will reduce anxiety and increase child cooperation during dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Dental anxiety
* Needs at least 2 dental treatment appointments

Exclusion Criteria:

* Medically compromised
* Cooperative, needs less than 2 dental treatment appointments

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Homeopathic Remedy First, Then Placebo: Homeopathic Remedy first, washout period and then Placebo
- Placebo First, Then Homeopathic Remedy: Placebo first, washout period and then Homeopathic Remedy
Period: First Intervention- 2 Days
Arm/Group | Homeopathic Remedy First, Then Placebo | Placebo First, Then Homeopathic Remedy
Started | 12 | 10
Completed | 6 | 5
Not Completed | 6 | 5
Period: Washout Period- 14 Days
Arm/Group | Homeopathic Remedy First, Then Placebo | Placebo First, Then Homeopathic Remedy
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention- 2 Days
Arm/Group | Homeopathic Remedy First, Then Placebo | Placebo First, Then Homeopathic Remedy
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Population: cross over design. Group 1 got homeopathic remedy on the first dental treatment, and placebo on the second treatment. Group 2 got placebo on the first dental treatment, homeopathic remedy on the second treatment
Arm/Group | All Study Population
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 7.09 [5 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 11

OUTCOME MEASURES:

1. Primary Outcome: Reducing Children's Anxiety
Description: Measuring levels of salivary cortisol and salivary α-amylase levels before dental treatment and after dental treatment .
Time Frame: Each dental apointment, aproximatly 30 minutes on the average
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Homeopathic Remedy: Group 1 got homeopathic remedy on the first dental treatment . Group 2 got homeopathic remedy on the second treatment.
- Placebo: Group 2 got placebo on the first dental treatment . Group 1 got placebo on the second treatment.
Arm/Group | Homeopathic Remedy | Placebo
Number analyzed (Participants) | 11 | 11
ng/ml
  cortisol pre treatment | 1.38 (1.45) | 2.28 (3.09)
  cortisol post treatment | 1.39 (2.9) | 4.37 (6.91)
  alpha amylase pre treatment | 56.02 (45.72) | 92.09 (110.65)
  alpha amylase post treatment | 76.82 (54.48) | 102.62 (104.42)

ADVERSE EVENTS:
Groups:
- Homeopathic Remedy: Cross over design. Group 1 got homeopathic remedy on the first dental treatment. Group 2 got homeopathic remedy on the second treatment.
- Placebo: Cross over design. Group 1 got placebo on the second dental treatment. Group 2 got placebo on the first treatment.
Arm/Group | Homeopathic Remedy | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes